CLINICAL TRIAL: NCT06464315
Title: Functional Substrate-Only Mapping Technique to Guide Ablation of Arrhythmogenic Substrate Underlying Ventricular Tachycardia
Brief Title: Functional Substrate-Only Guided VT Ablation
Acronym: NoMoVT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CARA-007-23F
Record Dates: First submitted 2024-05-23; First posted 2024-06-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Ventricular Tachycardia; Sudden Cardiac Death
Keywords: functional substrate mapping; conduction slowing; isochronal late activation mapping (ILAM); peak frequency signal analysis; deceleration zones
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac | interventions — X-Rays

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a prospective, single-blinded, randomized controlled trial comparing an experimental strategy of functional substrate mapping/ablation only without VT induction compared to standard VT mapping/ablation. The study subjects will be blinded to the randomization. The care providers doing the procedure (and/or investigators doing the procedure) cannot be blinded by nature of the intervention (either perform experimental mapping protocol or not).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Functional substrate mapping only without VT induction (Experimental): In this experimental arm, only functional substrate mapping will be used to guide ablation of conduction slowing regions, without VT induction or mapping during VT. Ablation targets of conduction slowing will be identified as: 1) deceleration zones of conduction slowing, previously defined as 3 isochrones coalescing within 1cm radius. 2) wavefront discontinuities represented by lines of conduction block, previously defined as late potentials with at least 20ms of isoelectric segment, and 3) regions of slow conduction characterized by high peak frequency (220-500Hz), which uses spectral frequency analysis to identify signals with highest frequency as a surrogate for slow conduction. All regions exhibiting any of these 3 surrogates of slow conduction will be ablated.
  Interventions: Procedure: Functional Substrate-Only Mapping without VT Induction
- Standard VT Mapping (Active Comparator): Standard-of-care mapping, including voltage mapping of intrinsic rhythm, entrainment, activation, and/or pace mapping, will be performed to guide VT ablation. Standard VT induction protocols will be performed.
  Interventions: Procedure: Standard-of-Care Mapping/Imaging

INTERVENTIONS:
Procedure: Functional Substrate-Only Mapping without VT Induction — In this arm, invasive maps will be constructed by annotating the latest deflection and peak frequency during voltage mapping of stable intrinsic rhythm to localize areas of slow conduction. Annotated algorithms are cleared by the FDA. No VT will be purposefully induced in this experimental arm.
  Other Names: Isochronal late activation mapping (ILAM), peak frequency analysis
  Arms: Functional substrate mapping only without VT induction
Procedure: Standard-of-Care Mapping/Imaging — Conventional invasive scar (voltage) and electrical VT (entrainment, activation, pace) mapping will be used to guide VT ablation. Functional substrate mapping will not be used in this arm. VT will be induced using standard protocols.
  Arms: Standard VT Mapping

SUMMARY:
Ventricular tachycardia (VT) is a leading cause of death and suffering in the Veteran population. Currently, ablation procedures are performed to destroy the diseased tissue that causes this problem. This study will test to see if an experimental strategy of only targeting regions of slow conduction without the induction of VT can improve the efficacy and safety of VT ablation. Once this study is completed, the investigators will know whether this ablation strategy could help increase the efficacy, safety and efficiency of ablation therapy of fatal heart rhythms.

DETAILED DESCRIPTION:
Ventricular tachycardia (VT) remains a leading cause of death and morbidity in the veteran population, but current ablation procedures to treat VT are limited by hemodynamic instability of induced VT during standard invasive activation mapping (up to 80% of induced VT), lengthy ablation procedures (~8 hours), and difficulty in accurately localizing the critical origination sites of VT. The long-term goal is to simplify VT ablation using invasive functional substrate mapping techniques to improve the safety, efficacy, and efficiency of VT catheter ablation. The overall objectives in this application are to i) perform a randomized clinical trial to test whether performing simplified VT ablation guided only by invasive functional substrate mapping without VT induction improves the safety and efficiency of VT ablation while maintaining similar efficacy compared to standard ablation and ii) mechanistically correlate abnormal functional substrate with VT origination sites localized using gold standard invasive activation mapping. The central hypothesis is that ablation of slowly conducting tissue characterized by high frequency signals is sufficient to eliminate VT and improves clinical outcomes of VT ablation. The rationale is that recently developed sophisticated techniques to characterize functionally abnormal tissue can localize critical VT-sustaining substrate without needing to subjecting patients to mapping of hemodynamically unstable VT which is routinely done during standard of care ablation. The central hypothesis will be tested by pursuing one primary specific aim: Perform a randomized clinical trial to determine whether VT ablation guided only by invasive functional substrate mapping without VT induction decreases procedure time, fluoroscopy time, and procedural complications while maintaining similar efficacy compared to standard VT ablation controls. This study also includes 2 sub-aims to uncover VT mechanisms characterizing the distance of slowly conducting tissue to VT exit sites and provide a method to unmask critical arrhythmogenic substrate in non-ischemic cardiomyopathy patients in whom scar is not easily identified. The research proposed is innovative because it tests a novel strategy using new algorithms that can identify the critical tissue sustaining VT without requiring the induction of VT. The proposed research is significant because a functional substrate-guided only approach to VT ablation while still localizing the critical tissue causing VT is expected to increase the safety, efficacy, and efficiency of treating a fatal heart rhythm disorder

ELIGIBILITY:
Inclusion Criteria:

* Men and women >18 years of age referred for clinically indicated VT ablation and experience monomorphic or polymorphic scar-based VT documented by telemetry, ICD interrogation, ECG or event monitoring.
* Scar-based VT is defined as VT in patients with structural heart disease (assessed with either abnormal nuclear perfusion imaging (>5% defect), late gadolinium uptake on cardiac MRI, wall thinning <10mm or calcified myocardium on cardiac CT, akinesis or hypokinesis on echocardiogram, presence of Q waves on ECG, history of myocardial infarct).
* Patients undergoing epicardial VT ablation and who undergo prophylactic percutaneous hemodynamic support devices will also be included.

Exclusion Criteria:

* Patients without structural heart disease will be excluded from the pri-mary analysis, but enrolled in a prospective registry
* Patients who are pregnant
* Presence of intracardiac thrombus
* active acute coronary ischemia with unrevascularized coronary artery disease (CAD >70% stenosis)
* Active bacteremia
* Inaccessible ventricles due to dual mechanical valves
* Inability to tolerate and inability to tolerate anticoagulation during ablation and for at least 1 month after ablation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2029-09-28 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to composite endpoint (VT recurrence, death, or acute hemodynamic decompensation) | 6 months
  Ventricular arrhythmia recurrence is defined by an episode of sustained VT lasting 30 seconds or appropriate implantable cardioverter-defibrillator therapy including anti-tachycardia pacing or shock.
  Acute hemodynamic decompensation is defined by escalation of at least 1 new high dose inotrope/pressor occurring after anesthesia induction with persistent requirement during stable rhythm, >20% drop in cardiac index, unplanned insertion of percutaneous hemodynamic support device.

SECONDARY OUTCOMES:
VT burden (ICD therapy including shocks and ATP, sustained VT episodes >30 seconds) | 6 months
  Total number of ICD therapies (ATP and shocks) and recorded sustained VT episodes>30 seconds, compared 6 months before and 6 months after ablation.
Total Mapping Time | immediately at the end of the procedure
  dwell time of multi-electrode mapping catheters
Total fluoroscopy time | immediately at the end of the procedure
  Total amount of fluoroscopy time during the entire procedure
total procedural time | immediately at the end of the procedure
  time from introduction of catheters to removal of catheters
Procedural adverse events or complications | 1 month
  Major complications include: new acute pericardial effusion requiring intervention, vascular complication requiring intervention, embolic stroke confirmed by brain imaging, limb ischemia requiring intervention, or bacteremia.
  Major adverse events include: cardiogenic shock (requiring escalation of inotropes or salvage mechanical circulatory support)
Use of general anesthesia | immediately at the end of the procedure
  Whether general anesthesia (intubation) is required/used during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Ho, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No